CLINICAL TRIAL: NCT00849134
Title: A First-Time-in-Human Randomised, Single Blind Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics, of Single Escalating Doses of GSK1482160, in Male and Female Healthy Subjects, and to Make a Preliminary Assessment of the Effect of Food.
Brief Title: First Time in Human Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and the Effect of Food of Single Assending Doses of GSK1482160.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111383
Record Dates: First submitted 2009-02-12; First posted 2009-02-23 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pain, Inflammatory
Keywords: First-Time-in-Human; Tolerability; Pharmacodynamics; Safety; Food Effect; Pharmacokinetics; Healthy Volunteers
MeSH Terms: conditions — Pain | interventions — N-(2-chloro-3-(trifluoromethyl)benzyl)-N-methyl-5-oxopyrrolidine-2-carboxamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1,2 & 3 (Placebo Comparator): This part of the study will start with a very low dose of study drug, which will then be gradually increased in subsequent doses. This is known as dose-rising and is the way to assess safety and tolerability (i.e. possible presence of any side effects that make taking the drug unpleasant) of increasing the study drug. Effects will be compared to those seen when a placebo is taken. Up to 3 groups of 8 healthy male and female volunteers may be enrolled.
  Interventions: Drug: GSK1482160 or placebo
- Cohort 4 (Active Comparator): If an investigation of food effect is not possible in Cohorts 2 or 3, this Cohort will be used to check if there is a difference in the blood levels of the study drug when taken with or without a high fat meal.
  Interventions: Drug: GSK1482160 or placebo

INTERVENTIONS:
Drug: GSK1482160 or placebo — GSK1482160 is a P2X7 receptor antagonist

SUMMARY:
This is a first-time-in-human study. The overall purpose of the study is to assess whether the drug is safe and well tolerated after single, increasing doses. At different doses, we will look to see how much of the drug gets into the bloodstream, how the drug is broken down and excreted and whether this is affected by the presence of food.

DETAILED DESCRIPTION:
GSK1482160 is a new drug to be developed for treating inflammatory pain (for example, arthritis). It acts on structures on inflammatory cells, known as P2X7 receptors. Blocking these receptors reduces the release of important inflammatory chemicals which exists within the body and are thought to play an important role in promoting inflammatory pain.

This study will start with a very low dose of study drug, which will then be gradually increased in subsequent doses. This is known as dose-rising and is the way to assess safety and tolerability (any side effects that make taking the drug unpleasant). Effects will be compared to those seen when a placebo (a "dummy" drug) is taken. Up to 4 groups of 8 healthy male or female volunteers will be enrolled into the study. In addition, part of the study will be used to check if there is a difference in the blood levels of the study drug when taken with or without a high fat meal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Male or female aged between 18 and 55 years inclusive.
3. A female subject is eligible to participate if she is of non-childbearing potential:
4. Non-childbearing potential is defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and oestradiol < 40 pg/ml (<140 pmol/L) is confirmatory.]1
5. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 5 x terminal half-lives after the last dose.
6. Body weight > 50 kg and BMI within the range 18.5 - 29.9 kg/m2 (inclusive).
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. The written informed consent form should be signed and dated.
8. QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block. A 12-lead ECG at pre-study screening, which in the opinion of the Principal Investigator or physician designee has no abnormalities that will compromise safety in this study. The specific inclusion criterion with regard to QT interval (either QTcb or QTcf, machine or manual over-read, males or females) is that QTc should be less than 450msec (based on single or average QTc of triplicate ECGs obtained over a brief recording period).
9. No abnormality on relevant clinical chemistry or haematology examination at the pre-study medical examination. Subjects with laboratory parameters outside the reference range for this age group will only be included if the principal Investigator or designee considers that such findings will not introduce additional risk factors. Consultation with the GSK medical monitor is required before such subjects may be included. In any case, liver function tests (including bilirubin, ALT, AST or alkaline phosphatase) and markers of renal function (including urea and creatinine) must be strictly within the normal range at screening.
10. Normal physical examination (providing no evidence of clinically active disease or physical or mental impairment). A subject with a clinical abnormality may be included only if the Principal Investigator or physician designee considers that the abnormality will not introduce additional risk factors and will not interfere with study procedures. Consultation with the GSK medical monitor is required before such subjects may be included.
11. A 24-hour Holter at pre-study screening, which in the opinion of the Principal investigator or physician designee has no abnormalities that will compromise safety in this study. If a rhythm abnormality is detected, the subject may be included in the study only if the Principle Investigator or physician designee considers that the abnormality will not introduce additional risk factors and will not interfere with study procedures. Consultation with Principal Investigator, GSK medical monitor and, if required, a specialist cardiologist will occur before such a subject may be included.

Exclusion Criteria:

1. The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
2. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
3. A positive test for HIV antibody.
4. Subjects with any risk factors for tuberculosis that include: (i) a history of either congenital or acquired immunosuppression (e.g. HIV), (ii) a history of any disorder that may be a function of altered immunomodulation (e.g. autoimmune disease), (iii) a history of any clinical condition or surgical procedure that places them at higher risk of TB (e.g. diabetes, sarcoidosis, gastrectomy and vagotomy, malignancy, leukaemia), (iv) a history of mycobacterial infection, including TB, (v) recent close contact (within the previous 48 months) with an individual known to be infected with TB, (vi) recent immigrants or residents (within the previous 48 months) from countries where TB is considered to be of high-prevalence. For the purposes of TB screening amongst applicants for UK visas, high prevalence countries include Bangladesh, Ghana, Burkina Faso, Cote d'Ivoire, Togo, Niger, Kenya, Eritrea, Somalia, Pakistan, Sudan, Tanzania, Thailand, Cambodia and Laos (http://www.ukvisasgov.uk/en/howtoapply/tbscreening).
5. History of regular excessive alcohol consumption within 6 months of the study defined as:
6. an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
8. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
9. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor that the medication will not interfere with the study procedures or compromise subject safety.ONFIDENTIAL HH2007/00234/
10. History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
11. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period before the screening visit.
12. Pregnant females as determined by positive serum hCG test at screening or urine hCG test prior to dosing.
13. Lactating females.
14. Females of child-bearing potential
15. Females receiving Hormone Replacement Theory
16. Unwillingness or inability to follow the procedures outlined in the protocol.
17. Urinary cotinine levels indicative of smoking or a history of regular use of tobaccoor nicotine-containing products within 6 months prior to screening.
18. Has a resting systolic blood pressure which is outside the range of 90 to 140 mmHg, diastolic blood pressure is outside the range of 50 to 90 mmHg or heart rate is outside the range 90 to 40 bpm.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2009-04-06 (Actual); Study Completion 2009-04-06 (Actual)

PRIMARY OUTCOMES:
Safety parameters, adverse events, change from baseline and number of subjects outside the normal range for blood pressure, heart rate, 12-lead electrocardiogram (ECG) and clinical laboratory parameters. | Throughout study
Levels of GSK1482160 and any breakdown products in the blood and urine. | Throughout study
Measuring the amount of inhibition of inflammatory chemical release from blood following dosing with GSK1482160. | Throughout study

SECONDARY OUTCOMES:
Levels of GSK1482160 and any breakdown products in the blood and urine when taken with and without food. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111383 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111383?search=study&study_ids=111383#rs
- Available data/document: Individual Participant Data Set: 111383 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111383 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111383 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111383 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111383 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111383 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111383 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register